CLINICAL TRIAL: NCT04122443
Title: A Randomized Study of Ibuprofen + Oxycodone/Acetaminophen Versus Ibuprofen + Acetaminophen for ED Patients With Insufficient Relief of Acute Musculoskeletal Pain After Treatment With Prescription Strength Ibuprofen
Brief Title: Acetaminophen (APAP) +/- Oxycodone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-10592
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Acetaminophen; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen (Active Comparator): Acetaminophen alone
  Interventions: Drug: Acetaminophen
- Oxycodone/ acetaminophen (Active Comparator): Oxycodone + acetaminophen
  Interventions: Drug: Acetaminophen; Drug: Oxycodone

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen 650mg
Drug: Oxycodone — Oxycodone 10mg
  Arms: Oxycodone/ acetaminophen

SUMMARY:
This is an emergency department based randomized study of oxycodone/ acetaminophen versus acetaminophen alone for patients with acute musculoskeletal pain refractory to ibuprofen

ELIGIBILITY:
Inclusion Criteria:

* Acute musculoskeletal pain: Any pain attributable to muscles, bones, joints, tendons, ligaments or supporting structures, as determined by the clinical team, of 10 days duration or less. Prior to the onset of acute pain, patients cannot have experienced pain in the same body region during the prior six months
* Pain has to be described as moderate or severe, when the patient is asked if the pain is mild, moderate or severe in intensity

Exclusion Criteria:

* Use of an non-steroidal anti-inflammatory drug within the previous six hours
* Use of acetaminophen within the previous six hours
* Use of an opioid within the previous ten days
* Chronic pain, defined as any pain on >50% of days for at least 3 months prior to onset of acute pain
* Gout

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 393 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment into Stage 1 (open label stage) commenced on December 2019 in two urban emergency departments in Bronx, NY. Enrollment was halted from March-June 2020 due to COVID-19, and then resumed and concluded October 2020.
Pre-assignment Details: During enrollment into Stage 1 (ibuprofen open label stage), 924 patients were screened for participation and 393 were enrolled. Of the 393, a total of 159 reported insufficient relief of pain from ibuprofen and requested more medication to treat the pain. Five patients who met criteria to progress to the randomized stage withdrew of their own volition. As such, 154 patients progressed to Stage 2. 77 were randomized to oxycodone/acetaminophen and 77 were randomized to acetaminophen alone.
Groups:
- Acetaminophen: Acetaminophen alone (Stage 2, Double blinded)
  Acetaminophen: Acetaminophen 650mg PO
- Oxycodone/Acetaminophen: Oxycodone + Acetaminophen (Stage 2, Double blinded)
  Acetaminophen: Acetaminophen 650mg PO
  Oxycodone: Oxycodone 10mg PO
- Ibuprofen: Ibuprofen - 600mg PO (Stage 1, Open label)
Period: Stage 1 - Open Label
Arm/Group | Acetaminophen | Oxycodone/Acetaminophen | Ibuprofen
Started | 0 | 0 | 393
Completed | 0 | 0 | 154
Not Completed | 0 | 0 | 239
Not completed — Satisfactory relief after ibuprofen administration. Exited study | 0 | 0 | 234
Not completed — Withdrawal by Subject | 0 | 0 | 5
Period: Stage 2 - Double Blinded
Arm/Group | Acetaminophen | Oxycodone/Acetaminophen | Ibuprofen
Started | 77 | 77 | 0
Completed | 77 | 77 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 393 patients were enrolled into Stage 1 (Ibuprofen open label stage). 154 patients progressed to Stage 2 (two-arm, double blinded) of the study. An analysis of baseline characteristics inclusive of only the 239 Stage 1 participants was not conducted. As such, Age, Sex/Gender, and Pain Assessment baseline data representing only Stage 1 participants is not available.
Groups:
- Ibuprofen + Acetaminophen: Acetaminophen alone (Stage 2, Double blinded)
  Acetaminophen: Acetaminophen 650mg PO
- Ibuprofen + Oxycodone/Acetaminophen: Oxycodone + Acetaminophen (Stage 2, Double blinded)
  Acetaminophen: Acetaminophen 650mg PO
  Oxycodone: Oxycodone 10mg PO
- Total: Total of all reporting groups
Arm/Group | Ibuprofen + Acetaminophen | Ibuprofen + Oxycodone/Acetaminophen | Total
Number analyzed (Participants) | 77 | 77 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (12) | 38 (13) | 37.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 40 | 76
  Male | 41 | 37 | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 77 | 77 | 393
Pain Assessment [Mean (Standard Deviation); unit: score on a scale] — Baseline Pain Assessment was determined using the Numeric Rating Scale (NRS) for evaluating pain. The rating was verbalized, and the subject was asked to estimate current pain intensity on an 11-point scale, where 0 indicated no pain at all and 10 indicated the worst imaginable pain. Higher scores were indicative of greater pain intensity.
  score on a scale | 8.2 (1.2) | 8.3 (1.3) | 8.3 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Assessment
Description: Stage 1 (Open label): No Outcome Measures assessed
  Stage 2 (Double blinded): Change in Pain Assessment from baseline was determined using the Numeric Rating Scale (NRS) for evaluating pain. The rating was verbalized, and the subject was asked to estimate current pain intensity on an 11-point scale, where 0 indicated no pain at all and 10 indicated the worst imaginable pain. Positive mean changes in NRS scores were associated with increased pain relief.
Time Frame: 2 hours following treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ibuprofen and Then Acetaminophen (Stage 2): Ibuprofen - 600mg PO (Stage 1, Open label)
  Acetaminophen alone (Stage 2, Double blinded)
  Acetaminophen: Acetaminophen 650mg PO
- Ibuprofen and Then Oxycodone/Acetaminophen (Stage 2): Ibuprofen - 600mg PO (Stage 1, Open label)
  Oxycodone + Acetaminophen (Stage 2, Double blinded)
  Acetaminophen: Acetaminophen 650mg PO
  Oxycodone: Oxycodone 10mg PO
Arm/Group | Ibuprofen and Then Acetaminophen (Stage 2) | Ibuprofen and Then Oxycodone/Acetaminophen (Stage 2)
Number analyzed (Participants) | 77 | 77
score on a scale | 2.9 (2.4) | 4.0 (2.6)
Statistical Analysis 1: Comparison: Ibuprofen and Then Acetaminophen (Stage 2) vs Ibuprofen and Then Oxycodone/Acetaminophen (Stage 2); Test type: Superiority; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [0.3 to 1.9]

2. Secondary Outcome: Sustained Pain Relief
Description: Stage 1 (Open label): No Outcome Measures assessed
  Stage 2 (Double blinded): Sustained pain relief was determined using a four-item ordinal scale. The rating was verbal and the subject was asked to describe their level of pain within two hours of medication administration and maintaining this level, without rescue medication, for 48 hours. The patients used the following descriptors: severe, moderate, mild, or none. For reporting responses of 'mild' and 'none' were aggregated into a single category and 'moderate' and severe' were aggregated into a separate category.
Time Frame: Up to 48 hours following medication administration
Measure: Number; unit: participants
Arm/Group | Ibuprofen and Then Acetaminophen (Stage 2) | Ibuprofen and Then Oxycodone/Acetaminophen (Stage 2)
Number analyzed (Participants) | 77 | 77
participants
  Mild/None | 33 | 43
  Moderate/Severe | 44 | 34
Statistical Analysis 1: Comparison: Ibuprofen and Then Acetaminophen (Stage 2) vs Ibuprofen and Then Oxycodone/Acetaminophen (Stage 2); Test type: Superiority; Mean Difference (Final Values) = 13, 95% CI 2-sided [-3 to 29]

3. Secondary Outcome: Adequacy of Analgesia
Description: Stage 1 (Open label): No Outcome Measures assessed
  Stage 2 (Double blinded): Adequacy of analgesia was determined by querying the participants by asking a single question: "Did the medication provided control your pain?" Answer choices: Yes (it did); No (It did not); and Unsure. The number of participants responses were summarized by category.
Time Frame: 2 hours following treatment
Population: Responses for 3 participants in the 'Acetaminophen' arm and 1 participant in the 'Oxycodone + Acetaminophen' arm were unavailable.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen and Then Acetaminophen (Stage 2) | Ibuprofen and Then Oxycodone/Acetaminophen (Stage 2)
Number analyzed (Participants) | 74 | 76
Participants
  Yes | 51 | 59
  No | 23 | 17
  Unsure | 0 | 0
Statistical Analysis 1: Comparison: Ibuprofen and Then Acetaminophen (Stage 2) vs Ibuprofen and Then Oxycodone/Acetaminophen (Stage 2); Test type: Superiority; Mean Difference (Final Values) = 9, 95% CI 2-sided [-5 to 23]

4. Secondary Outcome: Satisfaction With Medication
Description: Stage 1 (Open label): No Outcome Measures assessed
  Stage 2 (Double blinded): The number of participants demonstrating satisfaction with medication was determined by asking participants if the same medication regimen would be desired during a subsequent episode of pain. Possible responses included "Yes", "No" or "Unsure"
Time Frame: 2 hours following treatment
Population: Responses for 4 participants in the 'Acetaminophen' arm and 1 participant in the 'Oxycodone + Acetaminophen' arm were unavailable.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen and Then Acetaminophen (Stage 2) | Ibuprofen and Then Oxycodone/Acetaminophen (Stage 2)
Number analyzed (Participants) | 73 | 76
Participants
  Yes | 41 | 47
  No | 22 | 18
  Unsure | 10 | 11
Statistical Analysis 1: Comparison: Ibuprofen and Then Acetaminophen (Stage 2) vs Ibuprofen and Then Oxycodone/Acetaminophen (Stage 2); Test type: Superiority; Mean Difference (Final Values) = 6, 95% CI 2-sided [-10 to 21]

5. Secondary Outcome: Medication-related Adverse Events
Description: Stage 1 (Open label): No Outcome Measures assessed
  Stage 2 (Double blinded): The number of participants demonstrating medication-related adverse events was tabulated by treatment arm/group.
Time Frame: 2 hours following treatment
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen and Then Acetaminophen (Stage 2) | Ibuprofen and Then Oxycodone/Acetaminophen (Stage 2)
Number analyzed (Participants) | 74 | 76
Participants | 7 | 26

ADVERSE EVENTS:
Time Frame: Stage 1 (Open label) - Patients were not assessed for adverse events Stage 2 (Double blinded) - Up to 2 hours post treatment administration
Description: Stage 1 (Open label) - Patients were not assessed for adverse events
  Stage 2 (Double blinded) - Adverse event data was unavailable for 3 participants in the 'Acetaminophen' alone arm/group and 1 participant in the 'Oxycodone + Acetaminophen' arm/group.
Groups:
- Ibuprofen (Stage 1): Ibuprofen - 600mg PO (Stage 1, Open label)
Arm/Group | Ibuprofen and Then Acetaminophen (Stage 2) | Ibuprofen and Then Oxycodone/Acetaminophen (Stage 2) | Ibuprofen (Stage 1)
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/76 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/76 | 0/0
Other Adverse Events (participants affected / at risk) | 6/74 | 18/76 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibuprofen and Then Acetaminophen (Stage 2) (N=74) | Ibuprofen and Then Oxycodone/Acetaminophen (Stage 2) (N=76) | Ibuprofen (Stage 1) (N=0)
Dizziness (Nervous system disorders) | 2 | 6 | 0
Drowsiness (Nervous system disorders) | 6 | 17 | 0
Nausea (Gastrointestinal disorders) | 0 | 6 | 0
Nausea (Gastrointestinal disorders) | 0 | 5 | 0
Fatigue (General disorders) | 0 | 1 | 0
Itchiness (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Shakiness (Nervous system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT04122443/Prot_SAP_000.pdf